CLINICAL TRIAL: NCT04754113
Title: Effect of Prone Position on Lung Ventilation and Perfusion Matching in Non-intubated Patients With COVID-19 Pneumonia
Brief Title: Effect of Prone Position onV/Q Matching in Non-intubated Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 PPV
Record Dates: First submitted 2021-02-06; First posted 2021-02-15 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: COVID-19; prone position; ventilation and perfusion matching
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prone position (Experimental): patients from supine to prone for at least 3 hours than re-supine
  Interventions: Other: prone position

INTERVENTIONS:
Other: prone position — patient was helped into the prone position, patient received instructions of end expiratory occlusion lasting at least 10 seconds and, 1 seconds after the start, a bolus of 10 mL of 5% NaCl solution was injected via the central venous catheter

SUMMARY:
A prospective physiologic study, in participants with COVID-19-related pneumonia requiring supplemental oxygen (standard oxygen therapy or high-flow nasal cannula (HFNC)) less than 24 hours. The investigators assessed the effect of prone position on ventilation inhomogeneity and ventilation/perfusion mismatch by electrical impedance tomography (EIT).

DETAILED DESCRIPTION:
Once enrolled, an EIT dedicated belt containing 16 electrodes was placed around the participant's chest at the fifth or sixth intercostal space and connected it to an EIT monitor (PulmoVista 500; Dräger Medical GmbH, Lübeck, Germany).

Baseline data were collected during supine position (timepoint SP1), including demographic and anthropometric data, a baseline arterial blood gas measurement, and ventilation parameters including type of supplemental oxygen, respiratory rate, fractional concentration of oxygen in inspired air (FiO2). The participants received instructions of end expiratory occlusion lasting at least 10 seconds and, 1 seconds after the start, a bolus of 10 mL of 5% NaCl solution was injected via the central venous catheter. Subsequently, each participant was helped into the prone position and data collection，end expiratory occlusion and 10% NaCl solution injection were preformed again after approximately 30 min (timepoint PP1). The participant was then encouraged to maintain the prone position for at least 3 h before being helped back into the supine position. Clinical data collection, end expiratory occlusion and injection of a bolus of 10 mL of 5% NaCl solution were repeated again 1 h after resupination (timepoint SP2).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to75 years
2. admitted to intensive care unit with a confirmed diagnosis of COVID-19-related pneumonia
3. requiring supplemental oxygen (standard oxygen therapy or high-flow nasal cannula (HFNC)) less than 24 hours,
4. gave written or witnessed verbal informed consent.

Exclusion Criteria:

1. uncollaborative or had an altered mental status,
2. New York Heart Association class above II
3. history of severe chronic obstructive pulmonary disease
4. Contraindications to the use of EIT (e.g., presence of pacemaker or chest surgical wounds dressing) or prone position (as decided by the attending physician)
5. Impending intubation (on the basis of clinical judgment, including clinical and physiological parameters).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Ventilation-perfusion (V/Q) mismatch | prone position 1 hour
  V/Q mismatch was quantified as the percentage of pixels that were classified as ventilated but not perfused (dead space fraction) plus the percentage of those perfused but not ventilated (shunt fraction).
Ventilation-perfusion (V/Q) mismatch | resupination 1 hour
  V/Q mismatch was quantified as the percentage of pixels that were classified as ventilated but not perfused (dead space fraction) plus the percentage of those perfused but not ventilated (shunt fraction).

SECONDARY OUTCOMES:
Regional ventilation | Baseline，prone position 1hour, resupination 1 hour
  The percentage of relative pixel-level ventilation (Vpixel) distending dorsal lung regions at each study phase
regional perfusion | Baseline，prone position 1hour, resupination 1 hour
  The pixel-level relative regional pulmonary perfusion
The Global Inhomogeneity (GI) index | Baseline，prone position 1hour, resupination 1 hour
  higher values indicating less homogenous ventilation
PF raio | Baseline，prone position 1hour, resupination 1 hour
  PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, Study Director — Zhongda Hospital, School of Medicinr, Southeast Univerty
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Chao Y, Yuan X, Zhao Z, Frerichs I, Li Z, Sun Q, Chen D, Zhang R, Qiu H, Liu L. Physiologic effects of prone positioning on gas exchange and ventilation-perfusion matching in awake patients with AHRF. BMC Pulm Med. 2024 Dec 4;24(1):600. doi: 10.1186/s12890-024-03411-0. PMID 39663512